CLINICAL TRIAL: NCT00926887
Title: A Double-Blind, Randomized, Placebo-Controlled Evaluation of the Effect of the Erchonia(R) EML Laser on Reducing Pain Following Breast Augmentation Surgery
Brief Title: Low Level Laser Therapy to Reduce Pain After Breast Augmentation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBA-001
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Laser (Sham Comparator): Placebo Laser is an inactive light
  Interventions: Device: Placebo Laser
- Erchonia EML Laser (Active Comparator): Erchonia EML Laser uses two 7mW red 635nm wavelength light emitting CSRH Class IIIb laser diodes. The energy delivered is 1.5 J/cm2.
  Interventions: Device: Erchonia(R) EML Laser

INTERVENTIONS:
Device: Erchonia(R) EML Laser — Low level laser red light of 635 nm and delivering 1.5 joules/cm2.
  Arms: Erchonia EML Laser
Device: Placebo Laser — Inactive light
  Arms: Placebo Laser

SUMMARY:
The goal of the clinical study was to see if applying low level laser light therapy to the breasts during breast implant surgery could lessen pain experienced by 24 hours after the surgery.

DETAILED DESCRIPTION:
Substantial pain, discomfort and swelling following breast augmentation surgery is not uncommon. The ability of low level laser therapy to reduce swelling and inflammation that subsequently reduces pain has been well documented. This study aimed to evaluate the ability of low level laser therapy to reduce post-operative pain and swelling for individuals undergoing bilateral breast augmentation surgery, by 24 hours post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Suitability for breast augmentation surgery based on the need for correction of a congenital deformity or condition such as: Amastia, Hypomastia, Hypoplasia, Pectus Carinatum, Pectus Excavatum, OR a cosmetic breast enhancement indication, including: Augmentation to increase breast size, correction of ptotic (drooping) or pendulous (sagging) breasts, recontouring to obtain enhanced breast shape.
* Bilateral breast augmentation indication only.
* 18 to 55 years, inclusive.
* Female, only.
* Willingness, and ability, to refrain from consuming over-the-counter and/or prescription medications for the indication of the relief of pain and/or swelling, including any non-steroidal anit-inflammatory drugs (NSAIDs), from 48 hours immediately prior to the laser-assisted breast implant procedure through to one week post-procedure.

Exclusion Criteria:

* Breast augmentation procedures indicated for the purpose of breast reconstruction following mastectomy or an injury due to severe trauma.
* Presence of a specific connective tissue disorder.
* Inadequate tissue available to cover the implants.
* Consumption of any one or more of narcotics, opiates, and/or steroids.
* Inability to consume the following medications post-operatively due to allergy, intolerance, or any other reason:

  (i) Pain medication for the relief of post-operative pain of Lortab 10/500 or another drug within the combination narcotic analgesic drug category within which Lortab falls.

(ii) Antibiotic medication for reducing the risk of post-operative infection of Keflex 500 mg or Cipro 500 mg or another drug within the broad-spectrum antibiotic drug category within which Keflex and Cipro fall.

* Developmental disability or cognitive impairment that impacts a subject's ability to read and/or to understand the content of the informed consent form, and/or impacts a subject's ability to read and /or to understand and/or to complete the required case report form information for the clinical study.
* Significant psychological disorder(s) for which treatment has become necessary, including anxiety and depression; psychiatric hospitalization.
* Pregnancy or lactation.
* Prior surgery to the breast area, or to the area of the intended incision.
* Infection or wound in the intended areas of treatment.
* Involvement in litigation and/or receiving disability benefits related to the subject's breast(s).
* Participation in research over the preceding 90 days.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Jackson, MD, FACS, Principal Investigator; Gregory Roche, DO, Principal Investigator; Thomas L Jackson, MD, Principal Investigator

REFERENCES:
- See also: FDA 510(k)#K072206 clearance listing resulting from the outcome of this study — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=25548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 9/30/05 - 6/28/07 at private practice test site locations.
Pre-assignment Details: There were no significant events or approaches for the study following participant enrollment and prior to group assignment. All enrolled participants proceeded to group assignment.
Groups:
- Erchonia(R) EML Laser: The Erchonia(R) EML Laser uses two 7mw red 635nm wavelength light emitting CSRH Class IIIb laser diodes. The energy delivered is 1.5 J/cm2.
Period: Overall Study
Arm/Group | Placebo Laser | Erchonia(R) EML Laser
Started | 54 | 50
Completed | 54 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Laser | Erchonia(R) EML Laser | Total
Number analyzed (Participants) | 54 | 50 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 50 | 104
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 104
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Scored Less Than 30 on the 0-100 Visual Analog Scale (VAS)for Pain 24 Hours Post-operative.
Description: Self-reported Degree of Pain rating using the standardized 0-100 Visual Analog Scale (VAS) scale provided at 24 hours post-implant procedure, at which time the subject will not have taken any pain medication for at least four hours. The VAS ratings range from 0 to 100, where '0' represents 'no pain at all' and '100' represents 'worst pain imaginable.' A VAS of 30 is indicated as a cutoff threshold for 'success.' Participants who recorded a VAS rating of less than 30 were considered study 'successes' and are reported below.
Time Frame: 24 hours post-operative
Population: ITT Analysis with LOCF technique employed, as applicable.
Measure: Number; unit: participants
Arm/Group | Placebo Laser | Erchonia(R) EML Laser
Number analyzed (Participants) | 54 | 50
participants | 20 | 37
Statistical Analysis 1: Comparison: Placebo Laser vs Erchonia(R) EML Laser; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Swelling Evaluation Through Length by Width Breast Diameter Measurements
Time Frame: immediately, 24 hours & 7 days post surgery
Reporting Status: Not Posted

3. Secondary Outcome: Self-reported Degree of Pain Rating in the Breasts Area.
Time Frame: 24 hours, 7 days, 14 days & 28 days post surgery
Reporting Status: Not Posted

4. Secondary Outcome: Use of Pain Management Medication Post-surgically.
Description: Average number of rescue pain medication doses consumed across the 1st 7 post-operative days.
Time Frame: Through the 1st 7 post-operative days.
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: medication doses
Arm/Group | Placebo Laser | Erchonia(R) EML Laser
Number analyzed (Participants) | 54 | 50
medication doses | 20.26 (8.89) | 18.43 (10.03)
Statistical Analysis 1: Comparison: Placebo Laser vs Erchonia(R) EML Laser; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; t=-2.711; df=102; p<0.01

5. Secondary Outcome: Hydration Level Assessment
Time Frame: immediately, 24 hours & 7 days post surgery.
Reporting Status: Not Posted

6. Secondary Outcome: Infection Evaluation
Time Frame: 24 hours & 7 days post surgery
Reporting Status: Not Posted

7. Secondary Outcome: Wound Healing Evaluation According to the Modified Hollander Cosmesis Scale
Time Frame: 7 days post surgery
Reporting Status: Not Posted

8. Primary Outcome: Self-reported Pain Rating on the 0-100 VAS 24 Hours Post-operative.
Description: Self-reported Degree of Pain rating using the standardized 0-100 VAS scale provided at 24 hours post-implant procedure, at which time the subject will not have taken any pain medication for at least four hours. VAS values range from '0' representing 'no pain at all' to '100' representing 'worst pain imaginable.'
Time Frame: 24 hours
Population: Intention to treat (ITT) analysis with imputation technique of Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo Laser | Erchonia(R) EML Laser
Number analyzed (Participants) | 54 | 50
scores on a scale | 36.78 (24.62) | 21.40 (20.60)
Statistical Analysis 1: Comparison: Placebo Laser vs Erchonia(R) EML Laser; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; df=102, t=-3.44

ADVERSE EVENTS:
Arm/Group | Placebo Laser | Erchonia(R) EML Laser
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/50
Other Adverse Events (participants affected / at risk) | 0/54 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No